CLINICAL TRIAL: NCT00247923
Title: Endometrial Polyps. Pathophysiology and Clinical Consequences.
Brief Title: Endometrial Polyps: Pathophysiology and Clinical Consequences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP I/II/III; 22200205
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-02

CONDITIONS: Endometrial Polyp; Endometrial Cancer
Keywords: Endometrial polyps.; Angiogenesis.; Asymptomatic.; Symptoms.; Malignancy.; Treatment efficiency.; Vaginal bleeding.
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms; Uterine Hemorrhage

INTERVENTIONS:
Procedure: Hysteroscopic resection of endometrial polyps. (TCRP)

SUMMARY:
The aim of these studies is to study the natural history, the symptoms of, as well as the effect of hysteroscopic resection of endometrial polyps. Furthermore, another aim is to study new diagnostic techniques to differentiate between malignant and benign endometrial polyps.

DETAILED DESCRIPTION:
Study Part 1: New diagnostic methods for the prediction of malignancy in endometrial polyps: A prospective pilot study.

Study of angiogenesis by identification of specific angiogenesis factors in tissue biopsies from the endometrium and by Doppler ultrasound combined with IV contrast. We hope to find specific characteristics with new vessel formation in the endometrial polyp, which can play a role in the prognostic evaluation regarding the risk for cancer development. We will compare women with endometrial polyps and women with endometrial cancer to see if these methods of angiogenesis evaluation may be useful in separating benign polyps from premalignant and malignant polyps.

Study Part 2: The natural history of endometrial polyps. A prospective randomised study of patients with endometrial polyps.

Blood loss during menstruation is documented with the help of a standardized form (PBAC). The patients are randomized to hysteroscopic resection of the endometrial polyp or 6 months of observation. A new registration of blood loss during menstruation is performed by patients in both groups. In the intervention group, a new gynaecological examination 6 months after the resection documents the presence of residual polyp or symptoms. The other group is examined again after 6 months of observation. Symptoms and findings with the second examination are compared with symptoms and findings at the first examination, any changes are documented and the final outcome in the to groups are compared.

Study Part 3: The occurrence and natural history of asymptomatic endometrial polyps in perimenopausal women. A prospective controlled study.

Registration of blood loss during menstruation is documented with the help of a standardized form (PBAC) and gynaecological examination including SIS of 1000 randomly selected women in the age group 45-50. Where endometrial polyps are identified, we document the size and number of polyps and an endometrial biopsy is taken. After including a woman with an endometrial polyp in the study, the next woman without endometrial polyp is recruited to the control group. After one year, blood loss during menstruation is registered again, and all women with endometrial polyps as well as the control group have a new examination including vaginal ultrasound, SIS and endometrial biopsy. Symptoms and findings are compared with symptoms and findings at the first examination and all changes are documented. If the woman has a persistent endometrial polyp when examined at 1 year, she is offered treatment with hysteroscopic polyp resection.

ELIGIBILITY:
Inclusion Criteria:

* Study 1:

  * Endometrial polyp (EP) group: Presence of endometrial polyp verified by vaginal ultrasound examination.
  * Cancer group: Presence of endometrial cancer verified by histological examination.
* Study 2:

  * Pre- or perimenopausal women.
  * Presence of endometrial polyp verified by vaginal ultrasound.
* Study 3:

  * EP group: Presence of endometrial polyp verified by vaginal ultrasound.
  * Control group: Normal endometrium by vaginal ultrasound examination.

Exclusion Criteria:

* Study 1: Earlier severe allergic reactions.
* Study 2:

  * Postmenopausal patient.
  * Pregnancy.
  * Additional condition requiring treatment detected during examination. Malignancy or atypical hyperplasia detected by histological examination.
* Study 3:

  * Previous hysterectomy.
  * Pregnancy.
  * Additional condition requiring treatment detected during examination. Malignancy or atypical hyperplasia detected by histological examination.

Ages: 16 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1186 (Estimated)
Dates: Start 2005-10; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Study part 1. Angiogenesis factor levels in endometrial biopsies in patients with endometrial polyps compared to patients with endometrial cancer
Resistance in the feeding vessel measured by doppler examination combined with intravenous (i.v.) contrast in patients with endometrial polyps and endometrial cancer
Study part 2. Change in pictorial blood loss assessment chart (PBAC) score in intervention compared to observation group
Study part 3. Change in PBAC score in women with endometrial polyps compared to control group

SECONDARY OUTCOMES:
Associated factors for the development of endometrial polyps
Change in endometrial polyp size and symptoms after 6 and 12 months of observation

CONTACTS AND LOCATIONS:
Overall Officials: Olav Istre, MD., PhD., Principal Investigator — Department og Gynaecology, Ullevaal University Hospital, Oslo, Norway.
Locations (1):
- Gynaecologial department, Ullevaal University Hospital, Oslo, Oslo County, Norway